CLINICAL TRIAL: NCT06403176
Title: Arteriovenous Plasma Multiomics and Inflammatory Factors in Patients With Disorders of Consciousness
Brief Title: Arteriovenous Plasma Multiomics in Patients With Disorders of Consciousness
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: plasma multiomics
Record Dates: First submitted 2022-03-14; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2022-03

CONDITIONS: Disorders of Consciousness; Transient Ischemic Attack
Keywords: Plasma metabolism
MeSH Terms: conditions — Consciousness Disorders; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Plasma for metabolites and lipids
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Minimally conscious state (MCS): Minimally conscious state (MCS): have reproducible signs of awareness and exhibit fluctuations in consciousness
  Interventions: Other: No intervention
- Vegetative state (VS): Vegetative state (VS): can open their eyes and preserve sleep-wake cycles, but unaware of themselves and their surroundings
  Interventions: Other: No intervention
- Patients with In-Stent Restenosis: In-Stent Restenosis was defined as greater than 50% within or immediately adjacent (within 5 mm) to the stent implanted that was detected by digital subtraction angiography (DSA).
  Interventions: Other: No intervention
- Patients with Non-Restenosis: In-Stent Restenosis was defined as less than 50% within or immediately adjacent (within 5 mm) to the stent implanted that was detected by digital subtraction angiography (DSA).
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
In order to determine the abnormal cerebral metabolism in the pathological state, we compared the blood of internal jugular vein, superior vena cava and radial artery during central venous catheterization. Metabonomics, proteomics and inflammatory factor microarray were used to detect the material differences in arteriovenous blood of patients with disorders of consciousness. At the same time, we concurrently compared it with the peripheral plasma metabolome of two additional patient cohorts: those in-stent restenosis and non-restenosis.

DETAILED DESCRIPTION:
Background:It is unclear what substances the brain needs to ingest for its activity under pathological conditions

Method:The uptake and release of substances by the brain were observed by comparing arterial blood with internal jugular vein blood;The characteristics of brain metabolites were observed by comparing internal jugular vein blood with superior vena cava blood. Compared it with the peripheral plasma metabolome of two additional patient cohorts: those in-stent restenosis and non-restenosis.

Objective:By analyzing different substances, this paper briefly describes the pathological mechanism of patients with disorders of consciousness, and looks for potential prognostic biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1.Patients with consciousness disorder caused by various severe brain injuries

Exclusion Criteria:

1. Patients who have been judged brain dead
2. There are persistent epileptic activity, inhibition or seizure inhibition patterns
3. Recent fever, abnormal liver and kidney function
4. Previous history of neurological or mental illness
5. Have a history of tumor
6. Inflammatory bowel diseases, hyperlipidemia, gastritis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with consciousness disorder caused by various severe brain injuries were recruited at Intensive care unit of The First Affiliated Hospital of Zhejiang University and Intensive care unit of the Second Affiliated Hospital of Zhejiang University
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Patient clinical outcome | 12 months
  The patients were followed up for 12 months after blood collection to observe the clinical outcome

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No